CLINICAL TRIAL: NCT06650163
Title: Biologic Validation of Zr-89 Crefmirlimab Berdoxam CD8+ Minibody ImmunoPET in Human Brain Tumors
Brief Title: Zr-89 Crefmirlimab Berdoxam and Immuno-Positron Emission Tomography for the Imaging of Patients With Resectable Brain Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-000877; NCI-2024-08388 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-000877 (Other: UCLA / Jonsson Comprehensive Cancer Center); P30CA016042 (NIH); P50CA211015 (NIH); R01CA267726 (NIH)
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Glioma; Malignant Brain Neoplasm; Meningioma; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Glioma; Brain Neoplasms; Meningioma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Zr-89 crefmirlimab berdoxam + ImmunoPET) (Experimental): Patients receive Zr-89 crefmirlimab berdoxam IV over 5-10 minutes 3 days prior to scheduled surgical resection. Approximately 24 hours after receiving Zr-89 crefmirlimab berdoxam, patients undergo immuno-PET scans. Patients then undergo scheduled standard of care surgical resection of the brain tumor and brain biopsy. Additionally, patients undergo advanced physiologic and metabolic MRI and MRI prior to surgery.
  Interventions: Procedure: Advanced Magnetic Resonance Imaging; Procedure: Brain Surgery; Other: Electronic Health Record Review; Procedure: Immuno-Positron Emission Tomography Scan; Procedure: Magnetic Resonance Imaging; Procedure: Stereotactic Biopsy; Diagnostic Test: Zirconium Zr 89 Crefmirlimab Berdoxam

INTERVENTIONS:
Procedure: Advanced Magnetic Resonance Imaging — Undergo advanced MRI
  Other Names: AMRI
Procedure: Brain Surgery — Undergo brain surgery
Other: Electronic Health Record Review — Ancillary studies
Procedure: Immuno-Positron Emission Tomography Scan — Undergo immuno-PET
  Other Names: Immuno-PET Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Stereotactic Biopsy — Undergo stereotactic image-guided biopsy
Diagnostic Test: Zirconium Zr 89 Crefmirlimab Berdoxam — Undergo Zirconium Zr 89 Crefmirlimab Berdoxam PET
  Other Names: 89Zr-Crefmirlimab Berdoxam; 89Zr-Desferrioxamine-IAB22M2C; 89Zr-Df-Crefmirlimab; 89Zr-Df-IAB22M2C; Zirconium Zr 89-Df-Crefmirlimab; Zirconium Zr 89-Df-IAB22M2C; Zirconium Zr-89 Crefmirlimab Berdoxam

SUMMARY:
This phase I trial studies how well zirconium (Zr)-89 crefmirlimab berdoxam and immuno-positron emission tomography (PET) identifies areas of immune cell activity in patients with brain tumors that can be removed by surgery (resectable). One important predictor of the immune response is the presence and change in CD8 positive (+) tumor infiltrating lymphocytes (TIL) cells. Identifying the presence and changes in CD8+ cells can be challenging, particularly for participants with central nervous system (CNS) tumors, and usually requires invasive procedures such as repeat tissue biopsies, which may not accurately represent the immune status of the entire tumor. Zr-89 crefmirlimab berdoxam is known as a radioimmunoconjugate which consists of a radiolabeled anti-CD8+ minibody whose uptake can be imaged with PET. Upon administration, Zr 89 crefmirlimab berdoxam specifically targets and binds to the CD8+ cells. This enables PET imaging and may detect CD8+ T-cell distribution and activity and may help determine the patient's response to cancer immunotherapeutic agents more accurately. Giving Zr-89 crefmirlimab berdoxam along with undergoing immuno-PET imaging may work better at identifying immune cell activity in patients with resectable brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To verify the specificity of Zr-89 crefmirlimab berdoxam CD8+ minibody immunoPET in identifying regions of immune cell activity in human glioma patients using stereotactic image-guided biopsies and multiplexed immunohistochemistry (IHC).

EXPLORATORY OBJECTIVE:

I. To evaluate the associations between exploratory biomarkers, clinical outcomes, and adverse events which include:

Ia. Exploring whether changes in specific magnetic resonance imaging (MRI) parameters correlate with tumor and peripheral blood immune responses; Ib. Assessing the potential change in Zr-89 crefmirlimab berdoxam uptake in tumor tissue and correlation with CD8 infiltrate in tumor tissue; Ic. Explore the correlation of visual and semi-quantitative Zr-89 crefmirlimab berdoxam PET measurements with clinical outcome.

OUTLINE:

Patients receive Zr-89 crefmirlimab berdoxam intravenously (IV) over 5-10 minutes 3 days prior to scheduled surgical resection. Approximately 24 hours after receiving Zr-89 crefmirlimab berdoxam, patients undergo immuno-PET scans. Patients then undergo scheduled standard of care surgical resection of the brain tumor and brain biopsy. Additionally, patients undergo advanced physiologic and metabolic magnetic resonance imaging (MRI) and MRI prior to surgery on study.

After completion of study treatment, patients are followed up until death.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years of age
* Documentation of a diagnosis of brain tumor including brain metastases, any grade of gliomas and meningiomas
* The participant is scheduled for standard of care surgical tumor resection
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial

Exclusion Criteria:

* Male or female < 18 years of age
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Not medically cleared for surgery
* Individuals who cannot tolerate MRI scan or PET/CT scan
* Pregnant or breast-feeding women
* Serum creatinine OR measured or calculated creatinine clearance (Glomerular filtration rate [GFR] can be use in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X institutional upper limit of normal (ULN) OR >= 60mL/min for subjects with creatinine levels > 1.5 X institutional ULN

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin: =< 1.5 X institutional ULN OR direct bilirubin =< institutional ULN for subjects with total bilirubin levels > 1.5 institutional ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional ULN OR =< 5 X institutional ULN for subjects with Gilberts syndrome
* Albumin >= 2.5 mg/dL
* Patients with splenic dysfunction or post splenectomy
* Any abnormalities that would be a contraindication to gadolinium-based contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 month
  Analyses will be examined graphically and summarized by descriptive statistics. Data transformation may be applied to quantitative variables prior to analyses if deemed necessary.
Zirconium (Zr)-89 crefmirlimab berdoxam uptake | Up to 24 hours
  Will be determined by standardized uptake value-based quantitative measures relative to CD8+ tumor infiltrating lymphocytes density determined by immunohistochemistry from tumor biopsy samples. Analyses will be examined graphically and summarized by descriptive statistics. Data transformation may be applied to quantitative variables prior to analyses if deemed necessary. Will correlate immuno-positron emission tomography uptake with cytotoxic T-cell density across all tumor samples. Multivariate cox and log rank tests will be used to compare survival outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Prins, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States